CLINICAL TRIAL: NCT00000764
Title: Chemoprevention of Anal Neoplasia Arising Secondary to Anogenital Human Papillomavirus Infection in Persons With HIV Infection.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: ACTG 216; 11193 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Anus Neoplasms
Keywords: Interferon Alfa-2a; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Anus Neoplasms; Papillomavirus, Human; Papovaviridae Infections; Tumor Virus Infections; Isotretinoin
MeSH Terms: conditions — HIV Infections; Anus Neoplasms; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Tumor Virus Infections | interventions — Isotretinoin; Interferon alpha-2

INTERVENTIONS:
Drug: Isotretinoin
Drug: Interferon alfa-2a

SUMMARY:
PRIMARY: In Phase I, to define a broadly tolerable dose of isotretinoin that can be used in combination with interferon alfa-2a (IFN alfa-2a). In Phase II, to determine trends in efficacy of isotretinoin alone or in combination with IFN alfa-2a as chemoprevention (preventing progression or recurrence) of anal intraepithelial neoplasia ( AIN ) / squamous intraepithelial lesions ( SIL ) in patients with HIV infection.

SECONDARY: To evaluate the effects of isotretinoin alone or in combination with IFN alfa-2a on immune function markers, human papillomavirus (HPV) type, and HPV DNA levels.

Patients with HIV infection have a significant risk of recurrence following local ablation of intraepithelial neoplasia; thus, anogenital epithelial may become an increasingly important cause of morbidity, and possibly mortality, as the HIV epidemic matures. Clinical studies of non-HIV-infected subjects have established that synthetic retinoids inhibit the progression of epithelial preneoplastic conditions and some neoplastic states.

DETAILED DESCRIPTION:
Patients with HIV infection have a significant risk of recurrence following local ablation of intraepithelial neoplasia; thus, anogenital epithelial may become an increasingly important cause of morbidity, and possibly mortality, as the HIV epidemic matures. Clinical studies of non-HIV-infected subjects have established that synthetic retinoids inhibit the progression of epithelial preneoplastic conditions and some neoplastic states.

In the Phase I portion of the study, 20 patients per site each receive isotretinoin in escalating doses. If a patient experiences grade 2 or worse toxicity (or grade 3 or worse hypertriglyceridemia), dose is reduced to the previously tolerated dose for the remainder of the 6 week period. Patients are then reassessed for anal neoplasia; those with no progression and no grade 2 or worse toxicity receive an additional 6 weeks of isotretinoin in combination with interferon alfa-2a. For Phase II of the study, a separate group of patients who have undergone ablative therapy are randomized to one of three arms (26 patients/arm): isotretinoin alone at the dose tolerated by at least 60 percent of patients in Phase I; isotretinoin plus interferon alfa-2a; or observation only. Treatment continues for 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* PCP prophylaxis (required for patients with CD4 count < 200 cells/mm3).
* Chemoprophylaxis for candidiasis and herpes simplex.
* Metronidazole for up to 14 days.
* Erythropoietin.

Patients must have:

* HIV seropositivity.
* NO active opportunistic infection requiring treatment with prohibited drugs.
* Phase I - Current grade 1 AIN (i.e., low grade SIL) OR treated or untreated grade 2 or 3 AIN (i.e., high grade SIL).

Phase II - Prior histologically confirmed grade 2 or 3 AIN / high grade SIL, with ablative therapy within the past 30-90 days.

* Capability of complying with study protocol.

NOTE:

* The terms condyloma, grade 1 AIN, and low grade SIL are interchangeable. Grade 2 or 3 AIN is interchangeable with high grade SIL.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active medical problems for which the patient is undergoing evaluations or for which prohibited therapy is required.
* Other active malignancies requiring systemic therapy.
* Significant symptomatic cardiac disease.

NOTE:

* Patients with malignancies being managed with local therapy (e.g., Kaposi's sarcoma, basal cell carcinoma) may enroll at the discretion of the site investigator.

Concurrent Medication:

Excluded:

* G-CSF (filgrastim).
* Myelosuppressive antibiotics (except co-trimoxazole for PCP prophylaxis).
* Corticosteroids.
* Biologic response modifiers.
* Cytotoxic chemotherapy.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with the following prior conditions are excluded:

History of ventricular arrhythmias or myocardial infarction.

Prior Medication:

Excluded within 20 days prior to study entry:

* G-CSF (filgrastim).
* Myelosuppressive antibiotics (except co-trimoxazole for PCP prophylaxis).
* Corticosteroids.
* Biologic response modifiers.
* Cytotoxic chemotherapy.

Prior Treatment:

Excluded within 20 days prior to study entry:

* Radiation therapy.

Excluded within 14 days prior to study entry:

* Transfusion.

Active substance abuse or illegal drug use (alcohol consumption is strongly discouraged).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98
Dates: Study Completion 1996-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Palefsky JM, Study Chair; Northfelt DW, Study Chair; Kaplan LD, Study Chair; Critchlow C, Study Chair
Locations (1):
- University of Washington AIDS CRS, Seattle, Washington, United States